CLINICAL TRIAL: NCT01118962
Title: An Open-Label Extension Study to Assess the Safety and Seizure Frequency Associated With Long-Term Oral Lacosamide for Uncontrolled Primary Generalized Tonic-Clonic Seizures in Subjects With Idiopathic Generalized Epilepsy
Brief Title: Open-Label Extension Study to Assess the Safety and Seizure Frequency Associated With Lacosamide for Primary Generalized Tonic-Clonic Seizures in Subjects With Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0962; 2014-004375-23 (EudraCT Number)
Expanded Access: NCT03559673 (No longer available)
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Results first posted 2013-12-04 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-03

CONDITIONS: Epilepsy
Keywords: Primary Generalized Tonic-Clonic (PGTC) Seizures; Absence Seizures; Myoclonic Seizures; Idiopathic Generalized Epilepsy (IGE)
MeSH Terms: conditions — Epilepsy; Seizures; Epilepsy, Idiopathic Generalized | interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lacosamide (Experimental): Lacosamide was supplied as 50 mg and 100 mg tablets. The starting Lacosamide dose was the same dose reached by a subject at the end of SP0961 (NCT01118949).
  Lacosamide was administered twice daily (approx. 12 hours apart, once in the morning and once in the evening) in 2 equally divided doses.
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — Lacosamide was supplied as 50 mg and 100 mg tablets. The starting Lacosamide dose was the same dose reached by a subject at the end of SP0961 (NCT01118949). At the beginning of SP0962, the dose may be maintained, or increased or decreased by 100 mg /day, as deemed clinically appropriate to optimize tolerability and seizure reduction. Dose increases should be no faster than 100 mg/ day per week up to a maximum of 800 mg/ day. Lacosamide was administered twice daily (approx. 12 hours apart, once in the morning and once in the evening) in 2 equally divided doses for up to a 56-week Treatment Phase. The Treatment Phase was followed by a 5-week End-of-Study Phase, during which subjects had to be tapered off Lacosamide at a recommended decrease rate of 200 mg/ day per week.
  Other Names: Vimpat®

SUMMARY:
The purpose is to obtain data on the safety and seizure frequency associated with long-term oral Lacosamide for uncontrolled primary generalized tonic-clonic (PGTC) seizures in subjects with idiopathic generalized Epilepsy. Additionally, to allow subjects who have completed SP0961 (NCT01118949) to continue to receive Lacosamide.

ELIGIBILITY:
Inclusion Criteria:

* Subject completed the SP0961 (NCT01118949) study
* Subject is expected to benefit from participation in an open-label extension study with Lacosamide, in the opinion of the investigator

Exclusion Criteria:

* Subject meets the withdrawal criteria for SP0961 (NCT01118949) or is experiencing an ongoing Serious Adverse Event (SAE)

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (19):
- United States (19):
  - 603, Phoenix, Arizona
  - 602, Little Rock, Arkansas
  - 628, Aurora, Colorado
  - 613, Atlanta, Georgia
  - 617, Boise, Idaho
  - 614, Fort Wayne, Indiana
  - 605, Lexington, Kentucky
  - 616, Louisville, Kentucky
  - 619, Scarborough, Maine
  - 609, Bethesda, Maryland
  - 615, Chesterfield, Missouri
  - 607, New York, New York
  - 620, Columbus, Ohio
  - 608, Charleston, South Carolina
  - 601, Nashville, Tennessee
  - 612, Dallas, Texas
  - 610, Norfolk, Virginia
  - 623, Renton, Washington
  - 624, Madison, Wisconsin

REFERENCES:
- [Result] Wechsler RT, Yates SL, Messenheimer J, Leroy R, Beller C, Doty P. Lacosamide for uncontrolled primary generalized tonic-clonic seizures: An open-label pilot study with 59-week extension. Epilepsy Res. 2017 Feb;130:13-20. doi: 10.1016/j.eplepsyres.2016.12.015. Epub 2016 Dec 29. PMID 28086164
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study began enrollment in August 2010. The study completed in October 2012. The participant flow consists of the Safety Set (SS).
  The Safety Set consists of all subjects that were dosed at least once with Lacosamide (LCM).
Period: Overall Study
Arm/Group | Lacosamide
Started | 39
Completed | 29
Not Completed | 10
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 4
Not completed — Pregnancy | 1
Not completed — Non-compliance with Medicinal Product | 1

BASELINE CHARACTERISTICS:
Population: Baseline measurements consist of the Safety Set (SS).
  The Safety Set consists of all subjects that were dosed at least once with Lacosamide (LCM).
Arm/Group | Lacosamide
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 36
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 39
Weight [Mean (Standard Deviation); unit: Kilograms] | 77.66 (17.58)
Height [Mean (Standard Deviation); unit: Centimeters] | 167.88 (8.25)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) From Visit 1 to the End of Study (Approximately 61 Weeks)
Time Frame: From Visit 1 to the end of study (Approximately 61 weeks)
Population: Of the 39 subjects in the Safety Set (SS), 39 were included in this analysis.
  The SS consists of all subjects that were dosed at least once with Lacosamide (LCM).
Measure: Number; unit: participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 39
participants | 37

2. Primary Outcome: Number of Participants Withdrawn From the Study Due to Treatment-emergent Adverse Events (TEAEs) From Visit 1 to the End of Study (Approximately 61 Weeks)
Time Frame: From Visit 1 to the end of study (Approximately 61 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 39
participants | 2

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from August 2010 through October 2012. Adverse Event reporting consists of the Safety Set (SS). The Safety Set consists of all subjects that were dosed at least once with Lacosamide (LCM).
Arm/Group | Lacosamide
Serious Adverse Events (participants affected / at risk) | 3/39
Other Adverse Events (participants affected / at risk) | 35/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=39)
PNEUMONIA (Infections and infestations) | 1 (1)
CONVULSION (Nervous system disorders) | 1 (1)
MIGRAINE (Nervous system disorders) | 1 (1)
ABNORMAL BEHAVIOUR (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=39)
PALPITATIONS (Cardiac disorders) | 2 (2)
DIPLOPIA (Eye disorders) | 3 (4)
NAUSEA (Gastrointestinal disorders) | 5 (5)
DIARRHOEA (Gastrointestinal disorders) | 2 (2)
FATIGUE (General disorders) | 3 (4)
GAIT DISTURBANCE (General disorders) | 2 (2)
SEASONAL ALLERGY (Immune system disorders) | 3 (3)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 10 (13)
SINUSITIS (Infections and infestations) | 3 (3)
GASTROENTERITIS VIRAL (Infections and infestations) | 2 (3)
INFLUENZA (Infections and infestations) | 2 (2)
TOOTH ABSCESS (Infections and infestations) | 2 (2)
FALL (Injury, poisoning and procedural complications) | 4 (4)
JOINT SPRAIN (Injury, poisoning and procedural complications) | 4 (5)
CONTUSION (Injury, poisoning and procedural complications) | 3 (3)
EXCORIATION (Injury, poisoning and procedural complications) | 2 (2)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 2 (2)
SKIN LACERATION (Injury, poisoning and procedural complications) | 2 (2)
WEIGHT INCREASED (Investigations) | 4 (4)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2)
ARTERIAL BRUIT (Investigations) | 2 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 2 (2)
INCREASED APPETITE (Metabolism and nutrition disorders) | 2 (2)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (4)
DIZZINESS (Nervous system disorders) | 10 (12)
HEADACHE (Nervous system disorders) | 7 (12)
TREMOR (Nervous system disorders) | 6 (6)
POSTICTAL STATE (Nervous system disorders) | 2 (9)
ANXIETY (Psychiatric disorders) | 4 (5)
CONFUSIONAL STATE (Psychiatric disorders) | 4 (4)
DEPRESSION (Psychiatric disorders) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 (4)
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 2 (2)
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.